CLINICAL TRIAL: NCT07326449
Title: Measurement Of End-Tidal Carbon Dioxide Partial Pressure (PetCO2) Using A Portable Capnograph During Rest and Low-Loaded Steady State Work On An Ergometer: Test Of Reproducibility and Validation Against Standard Of Care Measurement During a Cardio Pulmonary Exercise Test.
Brief Title: Test-Retest Reliability And Validation For End-Tidal Carbon Dioxide Measurement (PetCO2) During Rest And Low-Loaded Steady State Work Using A Portable Capnograph.
Status: Enrolling by invitation | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Kristofer Hedman, MD, PhD, Senior Associate Professor, Linkoeping University
Other Study IDs: 2025-01777-01
Record Dates: First submitted 2025-12-17; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cardiopulmonary Exercise Test; End-Tidal Carbon Dioxide; VO2max; Ventilatory Physiology
Keywords: End-tidal carbon dioxide measurement; Ventilatory efficiency; Cardiopulmonary exercise test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1 - Healthy volunteers: Cohort 1 consists of 20 study participants eligable with the inclusion and exclusion criteria.

SUMMARY:
The goal of this observational study is to investigate exhaled carbon dioxide measuring during rest and low-loaded work using a portable device (capnograph) and standard of care apparatus during a cardiopulmonary exercise test (CPET) in healthy volunteers. The study aims to answer:

How reliable is exhaled end-tidal carbon dioxide measurement for an individual over time using both standard of care apparatus and a portable device during an ergometer test?

Do the measurements correlate between the portable device and standard of care apparatus?

How do changes in breathing instructions and placement of sampling cannula affect the measurements from the portable device (capnograph)?

How is the reliability over time of other well established values from a cardio pulmonary exercise test?

Participants will be asked to perform a modified cardiopulmonary exercise test on an ergometer twice, separated in time (1-4 weeks). Measurements are sampled alternating standard of care apparatus and a portable capnograph at rest and during low-loaded work.

DETAILED DESCRIPTION:
Study summery The study is an experimental methodological investigation involving research participants who are essentially healthy. Individuals who consent to participate and meet all inclusion criteria without any exclusion criteria will be eligible for the study.

Each participant will perform a modified maximal exercise test on an ergometer on two separate occasions (1 to 4 weeks). The ergospirometric exercise test will be performed on a ergometer (eBike Basic, GE Medical Systems, GmbH), with PetCO₂ measured at rest while seated on the bike and at various predetermined steady state levels during low to moderate loading. Participants will then continue the protocol with a ramping workload to maximal exertion. The test will be terminated when the participant no longer can maintain the pedaling cadence (60 rpm) or develops predefined abnormal symptoms.

Gas analysis will be conducted using breath-by-breath technology (Jaeger Oxycon Pro or Vyntus CPX; Viasys Healthcare) and the hand held monitor (Capnostream35, Medtronic) connected to the nasal cannula.

Two test leaders (medically trained, one of whom is a physician) will oversee the exercise test, with one managing the ergospirometric equipment and the other handling PetCO₂ measurement via the handheld monitor.

Data from the handheld capnograph will be recorded on a specially coded (study ID) protocol form. Ergospirometric data including symptom ratings will be stored in a patient database under the participant's personal identity number.

The exercise tests will be medically reviewed.

For data processing, coded protocol data from each participant will be compiled together with ergospirometric data in a dedicated database. Data will be handled in coded form, manually processed, and extrapolated for group-level analyses.

Additional information from the study protocol will include gender, age, height, and weight. Also, smoking habits, cardiovascular and pulmonary comorbidities and related medications, and any symptoms during exertion will be recorded.

Primary Research Question What is the reliability of PetCO₂ measurement in the same individual, using a handheld PetCO₂ monitor with nasal cannula compared to a closed respiratory gas analysis system (ergospirometry), during repeated measurements on two different days, at rest and at various levels of exertion during a cycle ergometer test?

Secondary Research Questions What is the agreement between PetCO₂ measured with a closed respiratory gas analysis system (ergospirometry) and a handheld PetCO₂ monitor with nasal cannula, at rest and during physical exercise at different exertion levels in a cycle ergometer test? For the handheld chandheld PetCO₂ monitor, how are the measured PetCO₂ values affected depending on whether sampling is done nasally or orally, and whether the subject is instructed to breathe freely or only through the nose or mouth? What is the reliability of other established measures obtained from ergospirometry, such as peak oxygen uptake and ventilatory efficiency, measured using the same ergospirometric equipment as in the questions above?

Hypotheses PetCO₂ values do not differ statistically significantly between two different measurement occasions at the same workload and measurement method, regardless of sampling method.

There is no systematic bias in PetCO₂ measurement with the handheld monitor compared to ergospirometric measurement at rest or during low to moderate intensity cycling.

There is no systematic bias due to different sampling methods of EtCO₂ using the handheld device.

Variation in PetCO₂ from both handheld and ergospirometry measurements is not clinically significantly greater than the variation in other established ergospirometric variables.

Sample Size The sample size was determined through an equivalence analysis for the primary research question, where the hypothesis is that the difference between two measurements (taken on two separate occasions at the same workload) falls within a clinically insignificant margin. The null hypothesis is that there is a clinically significant difference between the occasions.

A clinically relevant difference is defined as 0.1 kPa, with a standard deviation of the difference between occasions of 0.1 kPa, power of 80%, and significance level of 0.05. Based on these parameters, 16 participants are required. Accounting for an expected dropout rate of 20% , 20 participants will be recruited, corresponding to 40 completed exercise tests.

Statistical Methods Collected data on PetCO₂ are numerical and will be analyzed using parametric or non-parametric methods depending on the distribution. Descriptive analysis will be used to characterize the study population, presenting mean and standard deviation or alternatively median and interquartile range.

For reliability assessment, intraclass correlation coefficient (ICC) analysis will be performed. Additionally, the coefficient of variation (COV%) will be reported for each measurement. Bland-Altman analysis will be used to assess agreement with ergospirometric measurements, as well as to evaluate different sampling methods using the handheld device.

Missing Data Occasional missing values will not be imputed.

Outliers Apparent erroneous values, defined as values lying beyond 1.5 times the interquartile range below Q1 or above Q3, will be excluded during data processing.

Adverse events Any sensitive personal data, primarily concerning the individual's health, disclosed by a research participant may necessitate the study personnel to refer the individual to the appropriate healthcare provider.

The study is conducted within a regular hospital setting for exercise testing evaluation, with access to emergency medical expertise and equipment. Study personnel are licensed healthcare professionals with extensive experience and knowledge in managing acute, including life-threatening, medical conditions.

There is a possibility that unexpected findings or signs of illness may be identified during the exercise test. In such cases, the individual will be referred to the appropriate healthcare authority for further assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 70 years.
* Proficient in spoken and written Swedish.
* Capable of cycling on an exercise bicycle.

Exclusion Criteria:

* Current symptoms of upper respiratory tract infection or fever within the past 5 days
* Obesity (BMI > 30 kg/m²)
* Known respiratory pattern disorders/hyperventilation syndrome
* More than mild asthma or other pulmonary diseases
* Cardiovascular disease (except for hypertension with or without treatment, mild heart valve disease at most, previous pericarditis > 12 months prior)
* Known pregnancy
* Presence of exertion-related symptoms such as chest pain, dizziness, syncope, arrhythmia, or abnormal shortness of breath

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer research participants recruited through advertisements at the research group's workplaces.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Reliability of PetCO2 sampling repeated over time. | Up to 4 weeks
  Intra-class correlation coefficient and covariance for repeated measurements with the handheld capnopragh and ergospiromtry at the same workload over time.
  What is the reliability of PetCO₂ measurement in the same individual, using a handheld PetCO₂ monitor with mask/nasal cannula compared to a closed respiratory gas analysis system (ergospirometry), during repeated measurements on two different days, at rest and at various levels of exertion during a cycle ergometer test?

SECONDARY OUTCOMES:
Correlation of PetCO2 measurements between standard of care ergospirometry and handheld PetCO2 monitor | Up to 4 weeks
  Bland-Altman analysis of aggrement between PetCO₂ handheld device versus ergospirometric measurement with limits of agreement.
  What is the level of agreement between PetCO₂ measured with a closed respiratory gas analysis system (ergospirometry) and a handheld PetCO₂ monitor with mask/nasal cannula, at rest and during physical activity at different levels of exertion during a cycle ergometer test?
Correlation measured as agreement for different sampling methods on the handheld capnograph. | Up to 4 weeks
  Bland-Altman analysis for different sampling methods on the handheld capnograph. For the handheld carbon dioxide monitor, how are the measured PetCO₂ values affected depending on whether sampling of exhaled air is done nasally or orally, and whether the test subject is instructed to breathe freely or only through the nose?
Intraclass correlation coefficient and covariance for other established ergospirometric variables (VO2peak, VE/VCO2slope) | Up to 4 weeks
  Reliability over time of "well established" outcome variables from CPET (VO2peak, VE/VCO2slope, OUES, eqCO2nadir)

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer Hedman, PhD. Associate professor, Principal Investigator — Linkoeping University
Locations (1):
- Region Östergötland, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No